CLINICAL TRIAL: NCT06477419
Title: Phase 2 Study of Sacituzumab Govitecan-hziy in Patients With Previously Treated Mesothelioma
Brief Title: A Study of Sacituzumab Govitecan in People With Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-081
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mesothelioma; Mesotheliomas Pleural; Mesothelioma; Pleura
Keywords: Mesothelioma; Mesotheliomas Pleural; Mesothelioma; Pleura; Diffuse Pleural Mesothelioma; Sacituzumab; 24-081; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Mesothelioma (Experimental): Participants will have pathologically confirmed diffuse pleural mesothelioma. Patients will undergo cross-sectional imaging after the first 2 cycles and subsequently after every 3 cycles until disease progression. Biopsies will take place at screening, prior to cycle 3, and an optional biopsy at the end of treatment if consent was obtained and deemed to be safe and feasible. Patients treated on study who are removed prior to the Cycle 3 tumor assessment will be evaluated for toxicity only and replaced. All patients treated past the Cycle 3 tumor assessment will be include in the toxicity and efficacy assessments.
  Interventions: Drug: Sacituzumab govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab govitecan-hziy — After enrollment, participants will receive SG until disease progression or intolerable toxicity.

SUMMARY:
Participants will receive sacituzumab govitecan until their disease gets worse (progresses), they have severe side effects and cannot continue study treatment, or the participants or the study doctor thinks it's in your best interest to stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient, or legally authorized representative (LAR), willing and able to provide written informed consent for the trial
* Patient age ≥ 18 at time of consent
* Pathologically confirmed diffuse pleural mesothelioma
* Must have received at least one prior systemic therapy (platinum/pemetrexed, immunotherapy or a combination thereof)
* Measurable disease as defined primarily by the modified RECIST criteria for mesothelioma (at PI discretion RECIST v1.1 may be used)
* Consent to undergo a biopsy prior to Cycle 1 Day 1 and Cycle 3 Day 1 if deemed medically safe and feasible
* Eastern Cooperative Oncology Group (ECOG) score 0 or Karnofsky Performance Status ≥ 70%
* Adequate organ function, defined as

  * Absolute neutrophil count ≥ 1.5K/mcL
  * Platelet count ≥ 100K/mcL
  * Adequate renal function defined as creatinine clearance ≥ 30ml/min (as calculated by Cockcroft-Gault Formula)
  * Hemoglobin > 9g/dL (prior transfusion permitted if not within 7 days of enrollment)
  * Total bilirubin ≤1.5 x upper limit of normal (ULN) if no liver metastases or <3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases; subjects with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits
  * AST, ALT ≤ 2.5 x ULN (if liver metastases are present, ≤5 × ULN)
* If of childbearing potential, must be willing to use highly effective mode of contraception for at least one month prior, during, and for 2 months after the end of active therapy

Exclusion Criteria:

* Currently participating in another study and receiving another study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of the first dose of treatment
* Prior hypersensitivity to irinotecan or any components of sacituzumab govitecan-hziy
* Prior cytotoxic/immunologic systemic therapy within 3 weeks prior to study Day 1 or has not recovered (i.e., CTCAE v5 ≥ Grade 1 at baseline; from clinically significant adverse events due to a previously administered agent (excluding Grade 2 neuropathy)
* Known psychiatric or substance abuse disorders that would interfere with the requirements of the trial within the opinion of the investigator
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early stage prostate cancer, or in situ cervical cancer after definitive treatment
* Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg)

  o NOTE: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Patients who fit these criteria must use Hep B prophylaxis during treatment. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing
* Positive hepatitis C antibody (anti-HCV)

  o NOTE: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible
* Participant is positive for human immunodeficiency virus (HIV), with 1 or more of the following:

  * Receiving ART that may interfere with study treatment (consult sponsor for review of medication prior to enrollment)
  * CD4 count < 350 cells/mm3 at screening
  * AIDS-defining opportunistic infection within 6 months of start of screening
  * Not agreeing to start ART and be on ART > 4 weeks plus having HIV viral load <400 copies/mL at end of 4-week period (to ensure ART is tolerated and HIV controlled)
* Myocardial infarction, unstable angina, stroke, transient ischemic attack (TIA), or coronary/peripheral artery bypass graft, or any acute coronary syndrome within 6 months of start of study drug
* Congestive heart failure defined as New York Heart Association (NYHA) Class III-IV or hospitalization for congestive heart failure (any NYHA class) within 6 months of study Day 1
* Pregnant women or women who are breastfeeding or of childbearing potential and not using a highly effective method of birth control for at least one month prior to enrollment. If the risk of contraception exists, male and female subjects must use highly effective contraception throughout the study and for at least 60 days after last treatment. Highly effective contraception includes either 2 barrier methods (diaphragm, condom by the partner, copper intrauterine device, sponge, or spermicide), or 1 barrier method and 1 hormonal method (any oral, subcutaneous, intrauterine, or intramuscular registered and marketed contraceptive agent that contains an estrogen and/or a progesterone agent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2029-06-21 (Estimated); Study Completion 2029-06-21 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 2 years
  Clinical efficacy of Sacituzumab Govitecan/SG determined by overall response rate by modified (m)RECIST criteria v1.1. Overall response rate defined as participants who achieve complete response or partial response as best overall response by modified RECIST v1.1 criteria for mesothelioma.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Offin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org